CLINICAL TRIAL: NCT04417192
Title: A Pilot Study to Evaluate the Efficacy and Safety of Preoperative Olaparib Monotherapy and Preoperative Olaparib Plus Pembrolizumab Combination Therapy in Patients With HRD-Positive Stage III or IV Advanced Epithelial Ovarian/Fallopian Tube/Primary Peritoneal Cancer
Brief Title: Olaparib Monotherapy and Olaparib + Pembrolizumab Combination Therapy for Ovarian Cancer
Acronym: OLAPem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Toru Mukohara, Chief of Breast and Medical Oncology Division, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC1903
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This study has 2 cohorts. Cohort 1 is Olaparib monotherapy Cohort 2 is Olaparib plus Pembrolizumab combination therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib or Olaparib Plus Pembrolizumab (Experimental): Cohort 1 : Olaparib will be administered for 6 weeks before surgery. Cohort 2 : Olaparib and Pembrolizumab will be administered simultaneously for 2 cycles(6 weeks) before surgery.
  Interventions: Drug: Olaparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib will be administered at a dose of 300mg as oral dose, twice a day.
Drug: Pembrolizumab — Pembrolizumab will be administered at a dose of 200mg as a 30-minutes IV infusion, Q3W (25 minutes to 40 minutes are acceptable).

SUMMARY:
To evaluate the efficacy and safety of preoperative olaparib monotherapy and preoperative olaparib plus pembrolizumab combination therapy in patients with untreated stage III, IV high-grade serous or Grade 3 endometrioid ovarian cancer with Homologous Recombination Deficiency (HRD) positivity.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of preoperative olaparib monotherapy and preoperative olaparib plus pembrolizumab combination therapy in patients with untreated stage III, IV high-grade serous or Grade 3 endometrioid ovarian cancer with HRD positivity. The first cohort (Olaparib monotherapy : 10 cases) will be evaluated for the presence or absence of immune cell activation, and the tumor reduction effect will be evaluated in the second cohort (Olaparib plus pembrolizumab combination therapy : 20 cases).

ELIGIBILITY:
Inclusion Criteria:

1. Has given signed informed consent to participate in the clinical trial of her own will.
2. Is aged 20 years or older on the day of signing the informed consent.
3. Has been diagnosed with histologically confirmed, Stage III or IV epithelial ovarian, fallopian tube, or primary peritoneal cancer by the International Federation of Gynecology and Obstetrics (FIGO) staging system (2014), with a histological type of high-grade serous or Grade 3 endometrioid carcinoma.
4. Have measurable disease based on RECIST 1.1.
5. Is a candidate for debulking surgery.
6. Has an HRD-positive tumor.
7. Has an ECOG Performance Status of 0 or 1.
8. Laboratory test results within 21 days prior to enrollment have met the following organ function criteria. However, measurements within 14 days of blood transfusion or administration of granulocyte-colony stimulating factor (G-CSF) are excluded.

   * Neutrophil count ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min
   * T-Bil ≤ 2.0 mg/dL
   * ALT and AST ≤ 100 U/L (≤ 200 U/L if liver metastasis is present)
9. A woman of childbearing potential must agree to use contraception after signing the informed consent, throughout the study period, and until at least 120 days following the last dose of the study drug

Exclusion Criteria:

1. Has received previous allogeneic bone-marrow transplantation.
2. Has concurrent interstitial lung disease/pneumonitis, or a history of (noninfectious) interstitial lung disease/pneumonitis that required treatment with steroids. Interstitial lung disease/pneumonitis includes radiation pneumonitis.
3. Has received prior antitumor therapy (e.g., chemotherapy, molecular-targeted therapy, therapeutic antibody, endocrine therapy, immunotherapy, and investigational therapy).
4. Has received surgery under general anesthesia within 28 days prior to enrollment. However, surgery to diagnose ovarian/fallopian tube/peritoneal cancer performed under general anesthesia is allowed.
5. Has received radiation or radioactive isotope therapy within 28 days prior to enrollment.
6. Has uncontrolled pericardial effusion, pleural effusion, or peritoneal effusion.
7. Has a history of cerebral infarction, cerebral hemorrhage, or transient cerebral ischemia within 180 days prior to enrollment.
8. Has a history of deep vein thrombosis or pulmonary embolism.
9. Is receiving systemic glucocorticoid therapy or systemic immunosuppressive therapy.
10. Has a history of autoimmune disease.
11. Is infected with human immunodeficiency virus (HIV).
12. Is infected with active* hepatitis B or hepatitis C.

    *: Active hepatitis B is defined as HBs antigen positive.
13. Has a symptomatic infection within 14 days prior to enrollment.
14. Has received a live vaccine within 28 days prior to enrollment.
15. Has clinically critical cardiac disease (has a history of myocardial infarction or angina pectoris within 180 days prior to enrollment or has New York Heart Association [NYHA] class II or higher cardiac failure, uncontrolled arrhythmia, or QTc prolongation defined as QTc > 470 msec).
16. Has active brain metastasis or a tumor causing spinal cord compression.
17. Is pregnant or breastfeeding.
18. Has a history of severe allergy, anaphylaxis, or hypersensitivity induced by humanized chimeric antibodies.
19. Is allergic to biologics produced from Chinese hamster ovary (CHO) cells, carboplatin, or paclitaxel.
20. Has a known or suspected active malignancy that is different from the disease of interest in the clinical trial or has a history of other malignancy within 3 years prior to enrollment. However, cutaneous basal cell carcinoma and cervical carcinoma in situ are not part of this exclusion criterion.
21. Is unwilling to or unable to comply with the protocol.
22. Is not eligible to enroll in the clinical trial based on the judgment by the Investigator or Sub-investigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 weeks
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1.

SECONDARY OUTCOMES:
The incidence of adverse events | Up to 30 days after the last dose
  The incidences and types of adverse events that occur during treatment will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Chemotherapy response score (CRS) | 6 months from the end of registration
  To evaluate the effect of histopathological treatment on patients with serous carcinoma and metastasis to the omentum. The histopathological treatment effect is determined according to the chemotherapy response score (CRS)
Progression-free survival (PFS) | 6 months from the end of registration
  PFS is defined as the time from the first dose to the earlier of progression assessed by the Investigator per RECIST v. 1.1 (PD) or clinical criteria, or death due to any cause.
Overall survival (OS) | 6 months from the end of registration
  OS is defined as the time from the first dose to death due to any cause.

OTHER OUTCOMES:
Biomarkers | 2 years
  Relationship between the germline mutation and therapeutic effect
The change in tumor-infiltrating lymphocytes | 2 years
  Relationship between the change in tumor-infiltrating lymphocytes in tumor tissue before and after therapy, and the therapeutic effect
The therapeutic effect | 2 years
  Relationship between the Tumor Mutation Burden (TMB) and the therapeutic effect

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka